CLINICAL TRIAL: NCT04266392
Title: Molecular Imaging of Prostate Cancer Using Radiofluorinated PSMA Ligand
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Stony Brook University (Other)
Collaborators: Progenics Pharmaceuticals, Inc. (Industry)
Responsible Party: Principal Investigator, Dinko Franceschi, Clinical Associate Professor, Stony Brook University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 889520
Record Dates: First submitted 2020-02-10; First posted 2020-02-12 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-05

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: [18F]-DCFPyl Ligand

INTERVENTIONS:
Drug: [18F]-DCFPyl Ligand — To assess the performance of [18F]-DCFPyl PET with whole-body MRI and multiparametric pelvic/prostate MRI for PCa detection in men with recurrence as determined by biochemical PSA level or evidence on CIM. Results of tracer uptake and MRI image features on whole body PET/MRI and dedicated pelvic/prostate PET/MRI, alone and together, will be correlated and compared to detection of lesions on CIM that usually includes bone scan (BS) and CT scan of the abdomen and pelvis, or PET imaging with F-18 Fluciclovine.In addition, in patients who undergo biopsy when performed as standard of care, we will correlate image features directly with histopathological findings on lesion biopsy to directly demonstrate that 'radiotracer and/or MRI positive' lesions contain tumor cells.

SUMMARY:
Eligible patients have prostate cancer that was treated with surgery or radiation therapy for localized disease and there is evidence of biochemical recurrence and/or metastases on conventional imaging.The objective of this study is to assess the performance in detection of prostate cancer of a new positron emission tomography (PET) radiotracer for prostate cancer ([18F]-DCFPyl) combined with magnetic resonance imaging (MRI). Results of tracer uptake and MRI image features as whole body PET/MRI and dedicated pelvic/prostate PET/MRI, alone and together, will be correlated and compared to detection of lesions on conventional imaging modalities. Additionally, if the patient undergoes a biopsy as standard of care, image features will correlate directly with histopathological findings.Validation of this radiotracer can potentially lead to its use as a standard of care for future imaging and improve diagnosis and treatment guidance.This drug is not approved by the Food and Drug Administration (FDA) and is therefore considered experimental.There will be 20 subjects enrolled in this study; all of these patients will be enrolled at Stony Brook University Medical Center.

DETAILED DESCRIPTION:
The study objective is to assess the performance of [18F]-DCFPyl PET with whole-body MRI and multiparametric pelvic/prostate MRI for PCa detection in men with recurrence as determined by biochemical PSA level or evidence on CIM. Results of tracer uptake and MRI image features on whole body PET/MRI and dedicated pelvic/prostate PET/MRI, alone and together, will be correlated and compared to detection of lesions on CIM that usually includes bone scan (BS) and CT scan of the abdomen and pelvis, or PET imaging with F-18 Fluciclovine. In addition, in patients who undergo a biopsy when performed as standard of care, image features will correlate directly with histopathological findings on lesion biopsy to directly demonstrate that 'radiotracer and/or MRI positive' lesions contain tumor cells.

To test the hypothesis, this study is being proposed using the [18F]-DCFPyL PET tracer for the detection of PCa in patients with biochemical recurrence or evidence on CIM. The [18F]-DCFPyL PET tracer will be provided by the company Progenics Pharmaceuticals, Inc. (New York, New York) and conducted under an investigational new drug (IND) approval received by Stony Brook University.

ELIGIBILITY:
Inclusion Criteria:

* subject has prostate cancer treated with surgery, radiation therapy and/or chemotherapy for localized disease
* subject has biochemical recurrence defined in postsurgical patients as a PSA value = > 0.2 ng/mL followed by a subsequent confirmatory PSA value = >0.2 ng/mL according to the American Urological Association (AUA) guidelines, or three consecutive rises above the nadir in patients following radiation therapy according to the American Society for Radiation Therapy and Oncology (ASTRO).
* in most cases, it will be required that the patient has had a prior CIM scan (such as a BS, MRI, CT or PET with F-18 Fluciclovine) performed before enrollment in this study; the only exception would be if the PSA level of the patient is remarkably high indicating apparent recurrence.

Exclusion Criteria:

* less than 18 years of age (prostate cancer is not prevalent in the pediatric population);
* any contraindications to MRI imaging such as electrical implants, cardiac pacemakers or perfusion pumps;
* ferromagnetic implants such as aneurysm clips, surgical clips, prostheses, artificial hearts, valves with steel parts, metal fragments, shrapnel, tattoos near the eye, or ferromagnetic objects such as jewelry or metal clips in clothing;
* is unable to lie comfortably on a bed inside the scanner for 60 minutes as assessed by physical examination and medical history (e.g. back pain, arthritis);
* if they have had treatment with investigational drug within 30 days prior to trial enrollment;
* if they had administration of another radioisotope within five physical half-lives of trial enrollment;
* if they had radiation or chemotherapy within 4 weeks prior to trial enrollment;

Eligibility will be determined by a screening interview. All subjects recruited for the study will be able to withdraw from the study at any time.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-12-16 (Actual); Primary Completion 2021-10-15 (Actual); Study Completion 2021-10-15 (Actual)

PRIMARY OUTCOMES:
Comparison of PET PSMA and Conventional Imaging | Within 1 year from the PET Imaging study
  Compare [18F]DCFPyL PET imaging combined with whole body magnetic resonance imaging (MRI) and multiparametric pelvic/prostate MRI to conventional imaging modalities (CIM)--such as 99mTc-methylene diphosphonate bone scan (BS) and contrast-enhanced CT (CECT) of the abdomen and pelvis, or a newly approved PET imaging agent F-18 Fluciclovine, for the localization and determination of extent of recurrent/metastatic disease in patients with biochemical recurrence of prostate cancer or evidence of recurrence on CIM.
Sensitivity and Specificity of PET/MRI PSMA in biochemical recurrence | Within 1 year from the PET Imaging study
  Determine the sensitivity and specificity of [18F]-DCFPyL PET/MRI for extent of recurrent/metastatic disease in patients with biochemical recurrence.

CONTACTS AND LOCATIONS:
Overall Officials: Dinko Franceschi, MD, Principal Investigator — Stony Brook Cancer Center
Locations (1):
- Stony Brook University, Stony Brook, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rowe SP, Macura KJ, Ciarallo A, Mena E, Blackford A, Nadal R, Antonarakis ES, Eisenberger MA, Carducci MA, Ross AE, Kantoff PW, Holt DP, Dannals RF, Mease RC, Pomper MG, Cho SY. Comparison of Prostate-Specific Membrane Antigen-Based 18F-DCFBC PET/CT to Conventional Imaging Modalities for Detection of Hormone-Naive and Castration-Resistant Metastatic Prostate Cancer. J Nucl Med. 2016 Jan;57(1):46-53. doi: 10.2967/jnumed.115.163782. Epub 2015 Oct 22. PMID 26493203
- [Background] Szabo Z, Mena E, Rowe SP, Plyku D, Nidal R, Eisenberger MA, Antonarakis ES, Fan H, Dannals RF, Chen Y, Mease RC, Vranesic M, Bhatnagar A, Sgouros G, Cho SY, Pomper MG. Initial Evaluation of [(18)F]DCFPyL for Prostate-Specific Membrane Antigen (PSMA)-Targeted PET Imaging of Prostate Cancer. Mol Imaging Biol. 2015 Aug;17(4):565-74. doi: 10.1007/s11307-015-0850-8. PMID 25896814
- [Background] Chen Y, Pullambhatla M, Foss CA, Byun Y, Nimmagadda S, Senthamizhchelvan S, Sgouros G, Mease RC, Pomper MG. 2-(3-1-Carboxy-5-[(6-[18F]fluoro-pyridine-3-carbonyl)-amino]-pentyl-ureido)-pentanedioic acid, [18F]DCFPyL, a PSMA-based PET imaging agent for prostate cancer. Clin Cancer Res. 2011 Dec 15;17(24):7645-53. doi: 10.1158/1078-0432.CCR-11-1357. Epub 2011 Oct 31. PMID 22042970
- [Background] Dietlein M, Kobe C, Kuhnert G, Stockter S, Fischer T, Schomacker K, Schmidt M, Dietlein F, Zlatopolskiy BD, Krapf P, Richarz R, Neubauer S, Drzezga A, Neumaier B. Comparison of [(18)F]DCFPyL and [ (68)Ga]Ga-PSMA-HBED-CC for PSMA-PET Imaging in Patients with Relapsed Prostate Cancer. Mol Imaging Biol. 2015 Aug;17(4):575-84. doi: 10.1007/s11307-015-0866-0. PMID 26013479
- [Background] Tan H, Joseph D, Loh NK, McCarthy M, Leong E, Siew T, Segard T, Morandeau L, Trevenen M, Francis RJ. A pilot study of the utility of choline PET-CT in prostate cancer biochemical relapse following radical prostatectomy. J Med Imaging Radiat Oncol. 2016 Jun;60(3):374-81. doi: 10.1111/1754-9485.12455. Epub 2016 Apr 20. PMID 27094471
- [Background] O'Keefe DS, Bacich DJ, Heston WD. Comparative analysis of prostate-specific membrane antigen (PSMA) versus a prostate-specific membrane antigen-like gene. Prostate. 2004 Feb 1;58(2):200-10. doi: 10.1002/pros.10319. PMID 14716746
- [Background] Chang SS. Overview of prostate-specific membrane antigen. Rev Urol. 2004;6 Suppl 10(Suppl 10):S13-8. PMID 16985927
- [Background] Thompson IM, Valicenti RK, Albertsen P, Davis BJ, Goldenberg SL, Hahn C, Klein E, Michalski J, Roach M, Sartor O, Wolf JS Jr, Faraday MM. Adjuvant and salvage radiotherapy after prostatectomy: AUA/ASTRO Guideline. J Urol. 2013 Aug;190(2):441-9. doi: 10.1016/j.juro.2013.05.032. Epub 2013 May 21. PMID 23707439
- [Background] van der Pol CB, Schweitzer ME, Di Primio G, Sampaio ML, Kielar A, Clemons M, Jaberi A. Breast cancer and bone metastases: the association of axial skeleton MRI findings with skeletal-related events and survival. Breast Cancer Res Treat. 2014 Aug;146(3):583-9. doi: 10.1007/s10549-014-3046-z. Epub 2014 Jul 10. PMID 25007963
- [Background] Rowe SP, Macura KJ, Mena E, Blackford AL, Nadal R, Antonarakis ES, Eisenberger M, Carducci M, Fan H, Dannals RF, Chen Y, Mease RC, Szabo Z, Pomper MG, Cho SY. PSMA-Based [(18)F]DCFPyL PET/CT Is Superior to Conventional Imaging for Lesion Detection in Patients with Metastatic Prostate Cancer. Mol Imaging Biol. 2016 Jun;18(3):411-9. doi: 10.1007/s11307-016-0957-6. PMID 27080322